CLINICAL TRIAL: NCT02690701
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Effect of Secukinumab on Aortic Vascular Inflammation and Cardiometabolic Biomarkers After 12 Weeks of Treatment, Compared to Placebo, and up to 52 Weeks of Treatment With Secukinumab in Adult Subjects With Moderate to Severe Chronic Plaque-type Psoriasis
Brief Title: Study to Evaluate the Effect of Secukinumab Compared to Placebo on Aortic Vascular Inflammation in Subjects With Moderate to Severe Plaque Psoriasis
Acronym: VIP-S
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457AUS02
Record Dates: First submitted 2016-02-19; First posted 2016-02-24 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-07

CONDITIONS: Chronic Plaque Psoriasis
Keywords: psoriasis; plaque psoriasis; secukinumab; AIN457; biologic; monoclonal antibody; aortic vascular inflammation
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Secukinumab (Experimental): Eligible patients received secukinumab 300 mg once weekly at Baseline, Weeks 1, 2, 3 and 4 followed by monthly dosing starting at Week 8 through Week 48 inclusive
  Interventions: Drug: Secukinumab 300 mg
- Placebo then Secukinumab (Placebo Comparator): Eligible patients received placebo doses once weekly at Baseline, Weeks 1, 2, 3 and 4 followed by a dose after four weeks at Week 8.
  Beginning with the Week 12 dose, participants were switched to treatment with secukinumab 300 mg and were dosed once weekly at Weeks 12, 13, 14, 15 and 16 followed by monthly dosing through Week 48 inclusive.
  Interventions: Biological: Placebo

INTERVENTIONS:
Drug: Secukinumab 300 mg — Secukinumab 300 mg was provided in 1 mL prefilled syringes of 150 mg. Each dose of 300 mg secukinumab consisted of two secukinumab 150 mg injections once weekly for 5 weeks (Baseline, Weeks 1, 2, 3 and 4), followed by dosing every four weeks starting at Week 8 through Week 48 inclusive.
  The patients (or caregivers) self-injected each dose at the study site under the supervision of site personnel when injections occurred on days of study visits.
  The injections not occurring on days of study visits were done by the patients (or caregivers) at home.
  Other Names: AIN457 300 mg
  Arms: Secukinumab
Biological: Placebo — Placebo was provided in 1 mL prefilled syringe. Each placebo dose consisted of two placebo injections once weekly for five weeks (Baseline, Weeks 1, 2, 3, 4), then after four weeks at Week 8. At Week 12, patients were switched to receive 300 mg secukinumab once weekly for five weeks (Weeks 12, 13, 14, 15, 16) followed by monthly dosing through Week 48 inclusive.
  The patients (or caregivers) self-injected each dose at the study site under the supervision of site personnel when injections occured on days of study visits.
  The injections not occurring on days of study visits were done by the patients (or caregivers) at home.
  Arms: Placebo then Secukinumab

SUMMARY:
This study evaluated the effect of secukinumab compared to placebo on aortic vascular inflammation in adult patients who have moderate to severe plaque psoriasis that is poorly controlled by current psoriasis treatments.

ELIGIBILITY:
Inclusion Criteria:

- Males and females at least 18 years of age with moderate to severe plaque psoriasis

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque psoriasis
* Previous exposure to IL-17A or IL-17 receptor targeting agents.
* Other active or ongoing disease that may interfere with evaluation of psoriasis or places the patient at unacceptable risk
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2018-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Exton, Pennsylvania
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Gelfand JM, Shin DB, Duffin KC, Armstrong AW, Blauvelt A, Tyring SK, Menter A, Gottlieb S, Lockshin BN, Simpson EL, Kianifard F, Sarkar RP, Muscianisi E, Steadman J, Ahlman MA, Playford MP, Joshi AA, Dey AK, Werner TJ, Alavi A, Mehta NN. A Randomized Placebo-Controlled Trial of Secukinumab on Aortic Vascular Inflammation in Moderate-to-Severe Plaque Psoriasis (VIP-S). J Invest Dermatol. 2020 Sep;140(9):1784-1793.e2. doi: 10.1016/j.jid.2020.01.025. Epub 2020 Feb 21. PMID 32088207
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized Set consisted of all 91 participants who were randomly assigned to a treatment group
Groups:
- Secukinumab: Eligible participants received secukinumab 300 mg once weekly at Baseline, Weeks 1, 2, 3, and 4 followed by monthly dosing starting at Week 8 through Week 48
- Placebo: Eligible participants received placebo once weekly at Baseline, Weeks 1, 2, 3, and 4 followed by a dose after four weeks at Week 8; participants were switched to once weekly secukinumab 300 mg at Weeks 12, 13, 14, 15, and 16 followed by monthly dosing through Week 48
Period: Treatment Period 1
Arm/Group | Secukinumab | Placebo
Started (46) | 46 | 45
Completed (44) | 44 | 42
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment Period 2
Arm/Group | Secukinumab | Placebo
Started (44) | 44 (Completed Treatment Period 1 and continued to Treatment Period 2) | 42
Completed (41) | 41 (Completed Treatment Period 2) | 37
Not Completed | 3 | 5
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 39 | 80
  >=65 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 33 | 28 | 61
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 36 | 36 | 72
  Black | 1 | 3 | 4
  Asian | 6 | 2 | 8
  Other | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Aortic Vascular Inflammation as Measured by FDG-PET/CT
Description: Change from baseline in the target to background ratio from the whole aorta.
  Effect of secukinumab 300 mg subcutaneous (sc) compared to placebo on aortic vascular inflammation with respect to the change from baseline in the target (arterial vascular uptake) to background (venous blood pool) ratio from the aorta. The primary analysis time point was at Week 12.
  Increased aortic vascular inflammation as measured by (18F) fluorodeoxyglucose positron emission tomography with computer assisted tomography (FDG-PET/CT)
Time Frame: baseline, 12 weeks
Population: Full Analysis Set (FAS) included all participants assigned medication. Patients inappropriately randomized (eg, IRT was called in error for randomization of a screen failed patient) were excluded from this analysis set. Following intent-to-treat principle, participants were analyzed according to treatment they were assigned to at randomization
Measure: Mean (Standard Deviation); unit: target to background ratio (TBR)
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
target to background ratio (TBR)
  Baseline: number analyzed (Participants) | 43 | 42
  Baseline | 1.6615 (0.37380) | 1.6333 (0.33228)
  Change from Baseline at Week 12: number analyzed (Participants) | 43 | 42
  Change from Baseline at Week 12 | 0.0143 (0.25520) | 0.0655 (0.28086)
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Statistical analysis (Analysis of Covariance) of change from baseline in target to background ratio for regions of the aorta at Week 12 (Full Analysis Set); Test type: Superiority — This superiority trial compares secukinumab with placebo with a view of demonstrating the superiority of secukinumab over placebo with regards to a specific outcome measure; p = 0.3712, ANCOVA; Least Square Mean = -0.053, 95% CI 2-sided [-0.169 to 0.064], Standard Error of Mean 0.059

2. Secondary Outcome: Change in Adiponectin Total
Description: Change from baseline in Adiponectin to measure adiposity
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
ng/mL
  Baseline: number analyzed (Participants) | 44 | 42
  Baseline | 18799.0 (18608.48) | 19475.00 (18343.00)
  Change from Baseline at Week 12: number analyzed (Participants) | 44 | 42
  Change from Baseline at Week 12 | 1594.90 (15146.84) | -1076.40 (14565.60)

3. Secondary Outcome: Change in Apolipoprotein B
Description: Change from baseline in Apolipoprotein B levels, a marker predictive of diabetes
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
ng/mL
  Baseline: number analyzed (Participants) | 43 | 42
  Baseline | 0.1014 (0.04651) | 0.1033 (0.04451)
  Change from Baseline at Week 12: number analyzed (Participants) | 43 | 42
  Change from Baseline at Week 12 | 0.0020 (0.06331) | 0.0017 (0.04835)

4. Secondary Outcome: Change in CRP
Description: Change from baseline in C reactive protein (CRP), a measure of inflammation
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
mg/L
  Baseline: number analyzed (Participants) | 44 | 41
  Baseline | 6.1525 (8.23016) | 7.8676 (7.59860)
  Change from Baseline at Week 12: number analyzed (Participants) | 43 | 42
  Change from Baseline at Week 12 | -1.0016 (9.45281) | 1.1622 (15.84088)

5. Secondary Outcome: Change in Cholesterol
Description: Change from baseline in Cholesterol level
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
mg/dL
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 179.350 (30.01243) | 178.707 (38.92573)
  Change from Baseline at Week 12: number analyzed (Participants) | 43 | 42
  Change from Baseline at Week 12 | 10.6000 (30.27379) | -8.4878 (35.18247)

6. Secondary Outcome: Change in Fetuin A
Description: Change from baseline in Fetuin A, a marker predictive of diabetes
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
ng/mL
  Baseline: number analyzed (Participants) | 44 | 41
  Baseline | 988677.800781 (488494.3491043) | 1169947.724848 (79644.6884632)
  Change from Baseline at Week 12: number analyzed (Participants) | 44 | 41
  Change from Baseline at Week 12 | 90810.212003 (444791.4700461) | 45731.298018 (452743.5932412)

7. Secondary Outcome: Change in Ferritin
Description: Change from baseline in Ferritin, a marker predictive of diabetes
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
ng/mL
  Baseline: number analyzed (Participants) | 44 | 42
  Baseline | 111.953 (91.17931) | 122.040 (114.8715)
  Change from Baseline at Week 12: number analyzed (Participants) | 44 | 42
  Change from Baseline at Week 12 | -6.1006 (60.71995) | -17.118 (63.86703)

8. Secondary Outcome: Change in GlycA
Description: Change from baseline in glycoprotein acetylation (GlycA), a marker of inflammation
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
μmol/L
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 413.860 (65.34929) | 439.622 (60.44873)
  Change from Baseline at Week 12: number analyzed (Participants) | 40 | 41
  Change from Baseline at Week 12 | 0.5152 (59.46394) | -1.5420 (40.25958)

9. Secondary Outcome: Change in HDL Cholesterol
Description: Change from baseline in High Density Lipoprotein (HDL) Cholesterol, a cardiometabolic biomarker
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
mg/dL
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 43.3000 (10.20357) | 43.0732 (12.52276)
  Change from Baseline at Week 12: number analyzed (Participants) | 40 | 41
  Change from Baseline at Week 12 | -0.7500 (8.80195) | -1.1220 (8.10924)

10. Secondary Outcome: Change in HDL Function (Cholesterol Efflux)
Description: Change from baseline in High Density Lipoprotein (HDL) Cholesterol (cholesterol efflux) , a cardiometabolic biomarker
  Ratio of the pleated serum to removal of Cholesterol
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
ratio
  Baseline: number analyzed (Participants) | 41 | 41
  Baseline | 0.9535 (0.18986) | 1.0456 (0.17819)
  Change from Baseline at Week 12: number analyzed (Participants) | 41 | 41
  Change from Baseline at Week 12 | 0.1473 (0.23262) | 0.0541 (0.21902)

11. Secondary Outcome: HDL Particle Total
Description: Change from baseline in High Density Lipoprotein (HDL) Cholesterol Particle Total
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
μmol/L
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 29.2875 (5.38184) | 29.3634 (6.27442)
  Change from Baseline at Week 12: number analyzed (Participants) | 40 | 41
  Change from Baseline at Week 12 | -0.1375 (5.22900) | -0.1707 (5.12973)

12. Secondary Outcome: HDL Size
Description: Change from baseline in High Density Lipoprotein (HDL) Cholesterol size
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
nm
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 8.9350 (0.53280) | 8.9585 (0.56656)
  Change from Baseline at Week 12: number analyzed (Participants) | 40 | 41
  Change from Baseline at Week 12 | 0.0500 (0.47932) | 0.0073 (0.34161)

13. Secondary Outcome: HOMA-IR
Description: Homeostatic Model Assessment-Insulin Resistance (HOMA-IR) Insulin [uIU/mL (mU/L)] x Glucose (mg/dL) = HOMA-IR
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: HOMA-IR units
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
HOMA-IR units
  Baseline: number analyzed (Participants) | 44 | 42
  Baseline | 3.4901 (3.02479) | 5.5112 (6.22334)
  Change from Baseline at Week 12: number analyzed (Participants) | 44 | 42
  Change from Baseline at Week 12 | 0.9563 (2.23669) | -1.2764 (5.13505)

14. Secondary Outcome: Change in IL-2 Receptor A
Description: Interleukin-2 Receptor A (IL-2RA) is a marker predictive of diabetes
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
pg/mL
  Baseline: number analyzed (Participants) | 41 | 41
  Baseline | 25.5554 (59.47232) | 21.0665 (61.46295)
  Change from Baseline at Week 12: number analyzed (Participants) | 41 | 41
  Change from Baseline at Week 12 | -3.3606 (38.52458) | -1.1162 (6.31189)

15. Secondary Outcome: Change in IL-18
Description: Interleukin-18 (IL-18) is a marker predictive of diabetes
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
pg/mL
  Baseline: number analyzed (Participants) | 44 | 42
  Baseline | 1259.45 (1910.327) | 1308.47 (2454.672)
  Change from Baseline at Week 12: number analyzed (Participants) | 44 | 42
  Change from Baseline at Week 12 | 34555.1 (231199.6) | -627.77 (1874.377)

16. Secondary Outcome: Change in IL-6
Description: Interleukin 6 (IL-6) is a marker of inflammation
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
pg/mL
  Baseline: number analyzed (Participants) | 44 | 42
  Baseline | 5.6477 (20.81242) | 1.6658 (1.50954)
  Change from Baseline at Week 12: number analyzed (Participants) | 44 | 42
  Change from Baseline at Week 12 | 0.1334 (29.35524) | -0.0900 (1.78692)

17. Secondary Outcome: Change in Intermediate-Density Lipoprotein (IDL) Particle
Description: Intermediate-density lipoprotein (IDL) particle is a marker of cardiometabolic function
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: nmol/mL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
nmol/mL
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 284.350 (179.6482) | 271.049 (155.7413)
  Change from Baseline at Week 12: number analyzed (Participants) | 40 | 41
  Change from Baseline at Week 12 | 47.0500 (167.6253) | 2.3902 (160.6046)

18. Secondary Outcome: Change LDL Cholesterol
Description: Change from baseline in Low-Density Lipoprotein (LDL) Cholesterol as a marker of cardiometabolic function
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
mg/dL
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 122.475 (28.86040) | 121.049 (36.39708)
  Change from Baseline at Week 12: number analyzed (Participants) | 40 | 41
  Change from Baseline at Week 12 | 9.9750 (29.84532) | -6.2927 (34.42401)

19. Secondary Outcome: Change in Leptin
Description: Change from baseline in Leptin a marker of adiposity
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
pg/mL
  Baseline: number analyzed (Participants) | 44 | 42
  Baseline | 19913.4 (21835.66) | 36813.3 (62138.25)
  Change from Baseline at Week 12: number analyzed (Participants) | 44 | 42
  Change from Baseline at Week 12 | -1886.0 (11701.00) | -5595.9 (17042.08)

20. Secondary Outcome: LDL Particle Total
Description: Change from baseline in Low Density Lipoprotein (LDL) Cholesterol Particle Total
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
nmol/L
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 1236.35 (317.9542) | 1263.00 (447.3457)
  Change from Baseline at Week 12: number analyzed (Participants) | 43 | 42
  Change from Baseline at Week 12 | 114.250 (294.8695) | -111.39 (343.2109)

21. Secondary Outcome: LDL Size
Description: Change from baseline in Low Density Lipoprotein (LDL) Cholesterol size
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
nm
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 21.2200 (0.74977) | 21.1171 (0.76384)
  Change from Baseline at Week 12: number analyzed (Participants) | 40 | 41
  Change from Baseline at Week 12 | -0.0025 (0.70036) | 0.1439 (0.53807)

22. Secondary Outcome: Change in Triglycerides
Description: Triglycerides are a marker of cardiometabolic function
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
mg/dL
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 123.200 (52.90398) | 125.293 (79.10633)
  Change from Baseline at Week 12: number analyzed (Participants) | 40 | 41
  Change from Baseline at Week 12 | 11.5000 (62.56279) | -10.732 (60.25281)

23. Secondary Outcome: Change in TNF-α
Description: Change in Tumor necrosis factor (TNF, tumor necrosis factor alpha, TNFα is a marker of inflammation Also written as TNF-alpha
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
pg/mL
  Baseline: number analyzed (Participants) | 44 | 42
  Baseline | 2.3919 (1.79049) | 2.8089 (4.11492)
  Change from Baseline at Week 12: number analyzed (Participants) | 44 | 42
  Change from Baseline at Week 12 | -0.3577 (1.52948) | -0.9818 (3.85715)

24. Secondary Outcome: Change VLDL Particle Total
Description: Change in Very-low-density lipoprotein (VLDL) cholesterol level
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
nmol/L
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 52.9125 (26.92102) | 54.5829 (27.57024)
  Change from Baseline at Week 12: number analyzed (Participants) | 40 | 41
  Change from Baseline at Week 12 | 3.2500 (28.56421) | 3.2024 (25.40299)

25. Secondary Outcome: VLDL Size
Description: Change from baseline in Very Low Density Lipoprotein (VLDL) Cholesterol size
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
nm
  Baseline: number analyzed (Participants) | 40 | 41
  Baseline | 51.5650 (9.11152) | 50.1195 (9.51641)
  Change from Baseline at Week 12: number analyzed (Participants) | 40 | 41
  Change from Baseline at Week 12 | -0.3950 (9.30271) | -0.7927 (7.72572)

26. Secondary Outcome: Area and Severity Index 75 (PASI 75)
Description: Percentage of participants with PASI75 response (yes, no) PASI75 response = at least a 75% improvement (reduction) in PASI score compared to baseline
  Psoriasis Area and Severity Index ( PASI) is a tool for measuring the severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).
Time Frame: week 12
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
percentage of participants | 84.8 | 0.0

27. Secondary Outcome: Psoriasis Area and Severity Index 90 (PASI 90)
Description: Percentage of participants with PASI90 response (yes, no) PASI90 response = at least a 90& improvement (reduction) in PASI score compared to baseline
Time Frame: week 12
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
percentage of participants | 73.9 | 0.0

28. Secondary Outcome: Psoriasis Area and Severity Index 100 (PASI100)
Description: Percentage of participants with PASI100 response (yes, no) PASI100 response = complete clearing of psoriasis
Time Frame: week 12
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
percentage of participants | 37.0 | 0.0

29. Secondary Outcome: Investigator's Global Assessment Modified 2011 (IGA Mod 2011) Score of 0 or 1
Description: percentage of participants with IGA mod 2011 score of 0 or 1 (yes, no)
  Investigator's Global Assessment modified 2011 (IGA mod 2011) score of 0 or 1
  Statistical analysis (Cochran-Mantel-Haenszel test) of Novartis Investigator's Global Assessment Modified 2011 0 or 1 response by visit (Non-responder Imputation)
Time Frame: week 12
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
percentage of participants | 78.3 | 0.0

30. Secondary Outcome: Dermatology Life Quality Index (DLQI) Total Score
Description: Change from baseline in the DLQI total score
  Summary of analysis of change from baseline in DLQI at Week 12 and statistical analysis (using Analysis of Covariance) of change from baseline in DLQI at Week 12
  The higher the score, the more quality of life is impaired.
  0 - 1 no effect at all on patient's life 2 - 5 small effect on patient's life 6 - 10 moderate effect on patient's life 11 - 20 very large effect on patient's life 21 - 30 extremely large effect on patient's life
Time Frame: baseline, 12 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 46 | 45
scores on a scale
  Baseline | 12.30 (7.65) | 12.6 (7.21)
  Change from baseline at Week 12 | -9.4 (7.91) | -0.5 (3.97)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 48 weeks
Description: Arms/Groups cannot be provided for each intervention separately after week 12 because placebo participants were switched to secukinumab 300mg.
  Adverse Events were collected irrespective of intervention for the Placebo/Secukinumab 300 mg Arm/Group and it is not possible to determine which intervention each Adverse Event corresponded to
Groups:
- Secukinumab 300 mg: Secukinumab 300 mg
- Placebo/Secukinumab 300 mg: Placebo/Secukinumab 300 mg
- Total: Total
Arm/Group | Secukinumab 300 mg | Placebo/Secukinumab 300 mg | Total
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45 | 0/91
Serious Adverse Events (participants affected / at risk) | 5/46 | 0/45 | 5/91
Other Adverse Events (participants affected / at risk) | 21/46 | 18/45 | 39/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (N=46) | Placebo/Secukinumab 300 mg (N=45) | Total (N=91)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (N=46) | Placebo/Secukinumab 300 mg (N=45) | Total (N=91)
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 5
Bronchitis (Infections and infestations) | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 9 | 7 | 16
Sinusitis (Infections and infestations) | 0 | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 8
Dizziness (Nervous system disorders) | 1 | 3 | 4
Headache (Nervous system disorders) | 0 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT02690701/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT02690701/SAP_001.pdf